CLINICAL TRIAL: NCT04244435
Title: Consequences of Using Thoracic Epidural Analgesia for Coronary Artery Bypass Grafting
Brief Title: Neuroaxial Prophylaxis for CABG
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Volgograd State Medical University (Other)
Responsible Party: Principal Investigator, Mikhail I Turovets, MD, professor, Volgograd State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TEA-CABG
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Occlusion
Keywords: coronary artery bypass grafting; prevention of complication; neuroaxial prophylaxis; thoracic epidural analgesia
MeSH Terms: conditions — Coronary Occlusion | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic epidural analgesia (Experimental): CABG and thoracic epidural analgesia will be used for perioperative analgesia postoperative period
  Interventions: Procedure: CABG; Drug: thoracic epidural analgesia
- Opioids (Active Comparator): CABG and opioids will be used for perioperative analgesia
  Interventions: Procedure: CABG; Drug: analgesia of opioids
- CABG (Active Comparator): coronary artery bypass grafting with and without cardiopulmonary bypass
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — coronary artery bypass grafting with and without cardiopulmonary bypass
Drug: thoracic epidural analgesia — thoracic epidural analgesia at the level of 1-10 thoracic vertebrae (ropivacainum 0,2-0,5% 5-10 ml/h)
  Arms: Thoracic epidural analgesia
Drug: analgesia of opioids — Opioids will be used for perioperative analgesia
  Arms: Opioids

SUMMARY:
Investigators plan to study the effect of thoracic epidural analgesia on postoperative parameters (complication rate, duration of hospitalization, mortality, etc.) of coronary artery bypass grafting.

DETAILED DESCRIPTION:
Investigators plan to conduct a comparative analysis of early postoperative complications of coronary artery bypass grafting with and without cardiopulmonary bypass in patients with independent risk factors for the development of postoperative complications (advanced age, diabetes mellitus, chronic kidney disease, obesity, chronic obstructive pulmonary disease) with various types of anesthesiology benefits (general anesthesia and thoracic epidural analgesia versus general anesthesia and opioids). Investigators predict a decrease in the risk of developing cardiac, respiratory, infectious and renal complications, a reduction in the duration of intensive care, inpatient treatment and mortality.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery bypass grafting

Exclusion Criteria:

* Absolute contraindications for the use of thoracic epidural analgesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
hospital mortality | 1 year
Hospitalization duration | 1 year
Duration of treatment in the intensive care unit | up to 1 year

SECONDARY OUTCOMES:
Complications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital №1 of Volgograd State Medical University, Volgograd, Russia